CLINICAL TRIAL: NCT05499624
Title: Safety & Efficacy of Oral Mucosal Carbon Dioxide Pressure (POMCO2) Measurement to Monitor Tissue Perfusion
Brief Title: POMCO2 Clinical Study MicroTrend System pCO2 Sensor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in focus by the company.
Sponsor: ExoStat Medical, Inc. (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EXO-CL-5000
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Hypoperfusion
Keywords: Oral mucosal carbon dioxide pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MicroTrend System (Experimental): MicroTrend System is placed onto the subject's cheek and the subject will actively participate in the study for up to 6 hours, with up to 4 hours of sensor monitoring.
  Interventions: Device: MicroTrend System

INTERVENTIONS:
Device: MicroTrend System — The hands-free device measures oral mucosal carbon dioxide pressure (POMCO2) and functions outside of the body and does not require a surgical procedure or any significant deviation from standard practice to operate.

SUMMARY:
The objective of this non-significant risk (NSR) study is to evaluate the safety and efficacy of the MicroTrend System by correlating POMCO2 data with relevant clinical metrics including arterial pressure and heart rate.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-randomized, non-significant risk (NSR) study evaluating the safety and efficacy of the MicroTrend System, which is indicated for monitoring oral mucosal carbon dioxide pressure (POMCO2) in hospital patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized adult (age 22 years and older) in the critical care unit
2. Willing and able to provide independent written informed consent (or the patient's legal representative, if applicable)
3. Willing and physically able to comply with the study protocol and procedures

Exclusion Criteria:

1. Evidence of intra- or peri-oral, buccal, or gingival disease or trauma to the face or mouth that may interfere with MicroTrend System that is deemed clinically significant by the investigator
2. Any clinically significant medical health history or vital sign deemed by the investigator to potentially interfere with study conduct
3. Vulnerable subject populations (e.g., incarcerated or cognitively challenged adults)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Correlation between POMCO2 | 4-6 hours
  Assessed by the MicroTrend System and the relevant clinical metrics of mean arterial pressure and heart rate. Statistically significant correlations (defined as p < 0.05) will be deemed success for this purpose, with adjustment for multiplicity by the Hochberg-Holm method

CONTACTS AND LOCATIONS:
Overall Officials: Raul J Gazmuri, MD, PhD, Principal Investigator — Captain James A. Lovell Federal Health Care Center
Locations (1):
- Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois, United States